CLINICAL TRIAL: NCT01253187
Title: Open-label, Randomized, Three-fold Crossover Study to Investigate the Bioequivalence of Two Different Tablet Formulations Containing 0.02 mg Ethinylestradiol (EE) and 3 mg Drospirenone (DRSP) Without [SH T00186D] and With [SH T04532B] 0.451 mg L-mefolinate (Metafolin), and to Investigate the Bioequivalence of Two Different Tablet Formulations Containing 0.451 mg L-mefolinate (Metafolin) Without [SH T04532C] and With 0.02 mg EE/ 3 mg DRSP [SH T04532B] in 42 Healthy Young Women
Brief Title: Investigation of Bioequivalence of Ethinylestradiol (EE) and Drospirenone (DRSP) in Two Different Tablet Formulations: YAZ and YAZ + Levomefolate Calcium (Metafolin) & L-5-MTHF in Two Different Tablet Formulations: Levomefolate Calcium (Metafolin) and YAZ + Levomefolate Calcium (Metafolin)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Head Clinical Pharmacology, Bayer Healthcare AG
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 91460; 2005-003049-15 (EudraCT Number); 309664 (Other: Company Internal)
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Results first posted 2011-05-09 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Contraception
MeSH Terms: interventions — drospirenone; drospirenone and ethinyl estradiol combination; 5-methyltetrahydrofolate; levomefolate calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- EE 0.02 mg/DRSP 3 mg (YAZ, BAY86-5300) (Experimental): single oral administration of 1 film-coated SHT00186D tablet (YAZ), containing 0.020 mg ethinylestradiol (EE) + 3 mg drospirenone (DRSP)
  Interventions: Drug: EE 0.02 mg/DRSP 3 mg (YAZ, BAY86-5300)
- EE 0.02mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE20/DRSP/L-5-MTHF Ca) (Experimental): single oral administration of 1 film-coated SHT04532B tablet, containing 0.020 mg ethinylestradiol (EE) + 3 mg drospirenone (DRSP) + 0.451 mg Metafolin (L-5-methyltetrahydrofolate calcium [MTHF-Ca])
  Interventions: Drug: EE 0.02 mg/DRSP 3 mg/L-5-MTHF Ca 0.451 mg (EE20/DRSP/L-5-MTHF Ca)
- L-5-MTHF Ca 0.451 mg (Metafolin) (Experimental): single oral administration of 1 coated SHT04532C tablet, containing 0.451 mg Metafolin (L-5-methyltetrahydrofolate calcium [MTHF-Ca])
  Interventions: Drug: L-5-MTHF 0.451mg (Metafolin)

INTERVENTIONS:
Drug: EE 0.02 mg/DRSP 3 mg (YAZ, BAY86-5300) — Treatment group A: Single 1 film-coated tablet (Ethinylestradiol [EE] 0.02mg / Drospirenone [DRSP] 3mg) taken orally under fasting condition at intervals of at least one menstrual cycle.
  Arms: EE 0.02 mg/DRSP 3 mg (YAZ, BAY86-5300)
Drug: EE 0.02 mg/DRSP 3 mg/L-5-MTHF Ca 0.451 mg (EE20/DRSP/L-5-MTHF Ca) — Treatment group B: Single 1 film-coated tablet (Ethinylestradiol [EE] 0.02mg / Drospirenone [DRSP] 3mg / L-5-methyltetrahydrofolate [L-5-MTHF] 0.451mg) taken orally under fasting condition at intervals of at least one menstrual cycle.
  Arms: EE 0.02mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE20/DRSP/L-5-MTHF Ca)
Drug: L-5-MTHF 0.451mg (Metafolin) — Treatment group C: Single 1 coated tablet (L-5-methyltetrahydrofolate [L-5-MTHF] 0.451mg) taken orally under fasting condition at intervals of at least one menstrual cycle.
  Arms: L-5-MTHF Ca 0.451 mg (Metafolin)

SUMMARY:
The purpose of this study is examine and compare the uptake of YAZ (oral contraceptive containing drospirenone and ethinylestradiol) with or without levomefolate calcium (Metafolin, a registered vitamin supplement) in the body and to examine and compare the uptake of levomefolate calcium with or without YAZ in the body, in healthy volunteers not using hormonal contraception

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volunteer
* Age: 18 - 38 years inclusive
* Body mass index (BMI)1: ≥ 19 and < 28 kg/m²
* Regular cyclic menstrual periods at screening OR when using combined oral contraceptives during the recruitment period reporting of natural cyclic menstrual periods prior to their use
* Willingness to use non-hormonal methods of contraception during the complete trial OR previous tubal ligation

Exclusion Criteria:

* incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, excretion and effect of the study drugs will not be normal
* known or suspected sex-steroid influenced malignancies
* endometrial hyperplasia; genital bleeding of unknown origin; uterus myomatosus
* known or suspected tumors of the liver and pituitary
* presence or history of severe hepatic disease as long as liver function values have not returned to normal
* severe renal insufficiency or acute renal failure
* thrombophlebitis, venous / arterial thromboembolic diseases; presence or history of prodromi of a thrombosis
* other conditions that increase susceptibility to thromboembolic diseases
* known neuropsychiatric diseases, especially known or suspected epilepsy, and/ or deficient status of folate or vitamin B12
* use of any other medication within 2 cycles before first study drug administration which could affect the study aim
* use of potassium sparing drugs; use of folic acid containing supplements or medicines or use of any medication within 2 cycles before first study drug administration known to interfere with folate metabolism
* inadequate folate and/or Vitamin B12 status, clinically relevant deviations in red cell folate concentrations

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2006-10; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Dinox B.V., Groningen, Netherlands

REFERENCES:
- [Result] Blode H, Klipping C, Richard F, Trummer D, Rohde B, Diefenbach K. Bioequivalence study of an oral contraceptive containing ethinylestradiol/drospirenone/levomefolate calcium relative to ethinylestradiol/drospirenone and to levomefolate calcium alone. Contraception. 2012 Feb;85(2):177-84. doi: 10.1016/j.contraception.2011.05.015. Epub 2011 Jul 19. PMID 22067789

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy young women, aged 18 - 38 years inclusive, who were nonsmokers were enrolled from 20 October 2006 to 13 September 2007 at one center in Germany.
Pre-assignment Details: 77 female volunteers were screened according to the inclusion and exclusion criteria to determine that the volunteer was in a good state of health and appropriate for inclusion in the study, and 44 volunteers were randomized at one center.
Groups:
- Treatment Sequence A: YAZ, EE20/DRSP/L-5-MTHF Ca, Metafolin: YAZ for Period 1; EE20/DRSP/L-5-MTHF Ca for Period 2; Metafolin for Period 3. YAZ: single oral administration of 1 film-coated SHT00186D tablet (YAZ), containing 0.020 mg ethinylestradiol (EE) + 3 mg drospirenone (DRSP) / EE20/DRSP/L-5-MTHF Ca: single oral administration of 1 film-coated SHT04532B tablet, containing 0.020 mg ethinylestradiol (EE) + 3 mg drospirenone (DRSP) + 0.451 mg Metafolin (L-5-methyltetrahydrofolate calcium [MTHF-Ca]) / Metafolin: single oral administration of 1 coated SHT04532C tablet, containing 0.451 mg Metafolin (L-5-methyltetrahydrofolate calcium [MTHF-Ca]).
- Treatment Sequence B: YAZ, Metafolin, EE20/DRSP/L-5-MTHF Ca: YAZ for Period 1; Metafolin for Period 2; EE20/DRSP/L-5-MTHF Ca for Period 3. YAZ: single oral administration of 1 film-coated SHT00186D tablet (YAZ), containing 0.020 mg ethinylestradiol (EE) + 3 mg drospirenone (DRSP) / Metafolin: single oral administration of 1 coated SHT04532C tablet, containing 0.451 mg Metafolin (L-5-methyltetrahydrofolate calcium [MTHF-Ca]) / EE20/DRSP/L-5-MTHF Ca: single oral administration of 1 film-coated SHT04532B tablet, containing 0.020 mg ethinylestradiol (EE) + 3 mg drospirenone (DRSP) + 0.451 mg Metafolin (L-5-methyltetrahydrofolate calcium [MTHF-Ca]).
- Treatment Sequence C: EE20/DRSP/L-5-MTHF Ca, YAZ, Metafolin: EE20/DRSP/L-5-MTHF Ca for Period 1; YAZ for Period 2; Metafolin for Period 3. EE20/DRSP/L-5-MTHF Ca: single oral administration of 1 film-coated SHT04532B tablet, containing 0.020 mg ethinylestradiol (EE) + 3 mg drospirenone (DRSP) + 0.451 mg Metafolin (L-5-methyltetrahydrofolate calcium [MTHF-Ca]) / YAZ: single oral administration of 1 film-coated SHT00186D tablet (YAZ), containing 0.020 mg ethinylestradiol (EE) + 3 mg drospirenone (DRSP) / Metafolin: single oral administration of 1 coated SHT04532C tablet, containing 0.451 mg Metafolin (L-5-methyltetrahydrofolate calcium [MTHF-Ca]).
- Treatment Sequence D: EE20/DRSP/L-5-MTHF Ca, Metafolin, YAZ: EE20/DRSP/L-5-MTHF Ca for Period 1; Metafolin for Period 2; YAZ for Period 3. EE20/DRSP/L-5-MTHF Ca: single oral administration of 1 film-coated SHT04532B tablet, containing 0.020 mg ethinylestradiol (EE) + 3 mg drospirenone (DRSP) + 0.451 mg Metafolin (L-5-methyltetrahydrofolate calcium [MTHF-Ca]) / Metafolin: single oral administration of 1 coated SHT04532C tablet, containing 0.451 mg Metafolin (L-5-methyltetrahydrofolate calcium [MTHF-Ca]) / YAZ: single oral administration of 1 film-coated SHT00186D tablet (YAZ), containing 0.020 mg ethinylestradiol (EE) + 3 mg drospirenone (DRSP).
- Treatment Sequence E: Metafolin, YAZ, EE20/DRSP/L-5-MTHF Ca: Metafolin for Period 1; YAZ for Period 2; EE20/DRSP/L-5-MTHF Ca for Period 3. Metafolin: single oral administration of 1 coated SHT04532C tablet, containing 0.451 mg Metafolin (L-5-methyltetrahydrofolate calcium [MTHF-Ca]) / YAZ: single oral administration of 1 film-coated SHT00186D tablet (YAZ), containing 0.020 mg ethinylestradiol (EE) + 3 mg drospirenone (DRSP) / EE20/DRSP/L-5-MTHF Ca: single oral administration of 1 film-coated SHT04532B tablet, containing 0.020 mg ethinylestradiol (EE) + 3 mg drospirenone (DRSP) + 0.451 mg Metafolin (L-5-methyltetrahydrofolate calcium [MTHF-Ca]).
- Treatment Sequence F: Metafolin, EE20/DRSP/L-5-MTHF Ca, YAZ: Metafolin for Period 1; EE20/DRSP/L-5-MTHF Ca for Period 2; YAZ for Period 3. Metafolin: single oral administration of 1 coated SHT04532C tablet, containing 0.451 mg Metafolin (L-5-methyltetrahydrofolate calcium [MTHF-Ca]) / EE20/DRSP/L-5-MTHF Ca: single oral administration of 1 film-coated SHT04532B tablet, containing 0.020 mg ethinylestradiol (EE) + 3 mg drospirenone (DRSP) + 0.451 mg Metafolin (L-5-methyltetrahydrofolate calcium [MTHF-Ca]) / YAZ: single oral administration of 1 film-coated SHT00186D tablet (YAZ), containing 0.020 mg ethinylestradiol (EE) + 3 mg drospirenone (DRSP).
Period: Period 1
Arm/Group | Treatment Sequence A: YAZ, EE20/DRSP/L-5-MTHF Ca, Metafolin | Treatment Sequence B: YAZ, Metafolin, EE20/DRSP/L-5-MTHF Ca | Treatment Sequence C: EE20/DRSP/L-5-MTHF Ca, YAZ, Metafolin | Treatment Sequence D: EE20/DRSP/L-5-MTHF Ca, Metafolin, YAZ | Treatment Sequence E: Metafolin, YAZ, EE20/DRSP/L-5-MTHF Ca | Treatment Sequence F: Metafolin, EE20/DRSP/L-5-MTHF Ca, YAZ
Started | 7 | 8 | 7 | 7 | 9 | 6
Completed | 7 | 8 | 7 | 7 | 9 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Treatment Sequence A: YAZ, EE20/DRSP/L-5-MTHF Ca, Metafolin | Treatment Sequence B: YAZ, Metafolin, EE20/DRSP/L-5-MTHF Ca | Treatment Sequence C: EE20/DRSP/L-5-MTHF Ca, YAZ, Metafolin | Treatment Sequence D: EE20/DRSP/L-5-MTHF Ca, Metafolin, YAZ | Treatment Sequence E: Metafolin, YAZ, EE20/DRSP/L-5-MTHF Ca | Treatment Sequence F: Metafolin, EE20/DRSP/L-5-MTHF Ca, YAZ
Started | 7 | 8 | 7 | 7 | 9 | 6
Completed | 7 | 8 | 7 | 7 | 8 | 6
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Period: Period 3
Arm/Group | Treatment Sequence A: YAZ, EE20/DRSP/L-5-MTHF Ca, Metafolin | Treatment Sequence B: YAZ, Metafolin, EE20/DRSP/L-5-MTHF Ca | Treatment Sequence C: EE20/DRSP/L-5-MTHF Ca, YAZ, Metafolin | Treatment Sequence D: EE20/DRSP/L-5-MTHF Ca, Metafolin, YAZ | Treatment Sequence E: Metafolin, YAZ, EE20/DRSP/L-5-MTHF Ca | Treatment Sequence F: Metafolin, EE20/DRSP/L-5-MTHF Ca, YAZ
Started | 7 | 8 | 7 | 7 | 8 | 6
Completed | 6 | 7 | 7 | 7 | 7 | 6
Not Completed | 1 | 1 | 0 | 0 | 1 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0 | 0
Not completed — difficulty with blood sampling | 0 | 1 | 0 | 0 | 0 | 0
Not completed — non-compliance | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes all participants treated
Arm/Group | Entire Study Population
Number analyzed (Participants) | 44
Age Continuous [Mean (Standard Deviation); unit: Years] | 26.3 (6.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Maximum Concentration (Cmax) of EE Incl. Bioequivalence (BE) Evaluation
Description: Cmax refers to the highest measured drug concentration which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample
Time Frame: up to 96 hours after administration
Population: Note that not all samples were evaluable for each outcome measure. Therefore the number of participants analyzed not necessarily matches the number of completers.
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Groups:
- EE 0.02mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE20/DRSP/L-5-MTHF Ca): single oral administration of 1 film-coated SHT04532B tablet, containing 0.020 mg ethinylestradiol (EE) + 3 mg drospirenone (DRSP) + 0.451 mg Metafolin (L-5-methyltetrahydrofolate calcium [L-5-MTHF Ca])
Arm/Group | EE 0.02 mg/DRSP 3 mg (YAZ, BAY86-5300) | EE 0.02mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE20/DRSP/L-5-MTHF Ca)
Number analyzed (Participants) | 39 | 39
pg/mL | 39.6 [35.7 to 44.0] | 41.9 [37.6 to 46.7]
Statistical Analysis 1: Comparison: EE 0.02 mg/DRSP 3 mg (YAZ, BAY86-5300) vs EE 0.02mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE20/DRSP/L-5-MTHF Ca); 38 volunteers qualified for statistical analysis of BE whereas all 39 volunteers with valid concentration time profiles were included in the pharmacokinetic (PK) analysis; Test type: Non-Inferiority or Equivalence — A sample size of 6 volunteers per sequence was considered sufficient to establish bioequivalence, id est the 90%-confidence interval for the mean ratio is located completely within the equivalence interval limits of 80% and 125%; ANOVA — The equivalence test was done using a 90% confidence interval, no p-value was to be calculated; mean ratio = 106.03, 90% CI [98.86 to 113.72] — Point estimate for the ratio [(EE20/DRSP/L-5-MTHF Ca) / YAZ]. Bioequivalence is established if the 90% confidence interval fall within the equivalence interval limits of 80-125%

2. Primary Outcome: Mean Area Under the Concentration-time Curve From Administration to the Last Measurement [AUC(0-tlast)] of EE Incl. Bioequivalence (BE) Evaluation
Description: The AUC is a measure of systemic drug exposure, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample
Time Frame: up to 96 hours after administration
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pg·h/mL
Arm/Group | EE 0.02 mg/DRSP 3 mg (YAZ, BAY86-5300) | EE 0.02mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE20/DRSP/L-5-MTHF Ca)
Number analyzed (Participants) | 39 | 39
pg·h/mL | 358 [320 to 400] | 370 [332 to 412]
Statistical Analysis 1: Comparison: EE 0.02 mg/DRSP 3 mg (YAZ, BAY86-5300) vs EE 0.02mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE20/DRSP/L-5-MTHF Ca); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA — The equivalence test was done using a 90% confidence interval, no p-value was to be calculated; mean ratio = 103.47, 90% CI [99.16 to 107.98] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Mean Maximum Concentration (Cmax) of DRSP Incl. Bioequivalence (BE) Evaluation
Description: as for outcome 1
Time Frame: up to 168 hours after administration
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | EE 0.02 mg/DRSP 3 mg (YAZ, BAY86-5300) | EE 0.02mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE20/DRSP/L-5-MTHF Ca)
Number analyzed (Participants) | 35 | 36
ng/mL | 25.4 [23.3 to 27.7] | 26.7 [24.5 to 29.1]
Statistical Analysis 1: Comparison: EE 0.02 mg/DRSP 3 mg (YAZ, BAY86-5300) vs EE 0.02mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE20/DRSP/L-5-MTHF Ca); 33 volunteers qualified for statistical analysis of BE whereas all 35 (YAZ) and 36 (EE20/DRSP/L-5-MTHF Ca) volunteers with valid concentration time profiles were included in the pharmacokinetic (PK) analysis; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA — The equivalence test was done using a 90% confidence interval, no p-value was to be calculated; mean ratio = 105.24, 90% CI [97.30 to 113.83] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Mean Area Under the Concentration-time Curve From Administration to the Last Measurement [AUC(0-tlast)] of DRSP Incl. Bioequivalence (BE) Evaluation
Description: as for outcome 2
Time Frame: up to 168 hours after administration
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng·h/mL
Arm/Group | EE 0.02 mg/DRSP 3 mg (YAZ, BAY86-5300) | EE 0.02mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE20/DRSP/L-5-MTHF Ca)
Number analyzed (Participants) | 35 | 36
ng·h/mL | 386 [352 to 424] | 383 [346 to 424]
Statistical Analysis 1: Comparison: EE 0.02 mg/DRSP 3 mg (YAZ, BAY86-5300) vs EE 0.02mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE20/DRSP/L-5-MTHF Ca); [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA — The equivalence test was done using a 90% confidence interval, no p-value was to be calculated; mean ratio = 100.48, 90% CI [97.28 to 103.79] — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: Mean Maximum Concentration (Cmax) of L-5-methyl-THF (Baseline Corrected) Incl. Bioequivalence (BE) Evaluation
Description: The baseline corrected Cmax is a measure of the highest measured drug concentration provided solely by the treatment after subtracting endogenous L-5-methyl-THF level. It is obtained by collecting a series of blood samples, measuring the concentrations of L-5-methyl-THF in each sample and by subtracting the pre-treatment concentration.
Time Frame: up to 12 hours after administration
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: nmol/L
Groups:
- L-5-MTHF Ca 0.451 mg (Metafolin): single oral administration of 1 coated SHT04532C tablet, containing 0.451 mg Metafolin (L-5-methyltetrahydrofolate calcium) [L-5-MTHF Ca]
Arm/Group | EE 0.02mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE20/DRSP/L-5-MTHF Ca) | L-5-MTHF Ca 0.451 mg (Metafolin)
Number analyzed (Participants) | 39 | 40
nmol/L | 44.3 [40.0 to 49.2] | 44.2 [39.1 to 49.9]
Statistical Analysis 1: Comparison: EE 0.02mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE20/DRSP/L-5-MTHF Ca) vs L-5-MTHF Ca 0.451 mg (Metafolin); 39 volunteers qualified for statistical analysis of BE whereas all 39 (EE20/DRSP/L-5-MTHF Ca) and 40 (Metafolin) volunteers with valid concentration time profiles were included in the pharmacokinetic (PK) analysis; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA — The equivalence test was done using a 90% confidence interval, no p-value was to be calculated; mean ratio = 99.88, 90% CI [91.24 to 109.34] — Point estimate for the ratio [(EE20/DRSP/L-5-MTHF Ca) / Metafolin]. Bioequivalence is established if the 90% confidence interval fall within the equivalence interval limits of 80-125%

6. Primary Outcome: Mean Area Under the Concentration-time Curve From Administration to the Last Measurement [AUC(0-tlast)] of L-5-methyl-THF (Baseline Corrected) Incl. Bioequivalence (BE) Evaluation
Description: The baseline corrected AUC is a measure of the systemic drug exposure provided by the treatment excluding the endogenous L-5-methyl-THF level. It is obtained by collecting a series of blood samples, measuring the concentrations of L-5-methyl-THF in each sample and by subtracting the pre-treatment concentration.
Time Frame: up to 12 hours after administration
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: nmol·h/L
Groups:
- L-5-MTHF Ca 0.451 mg (Metafolin): single oral administration of 1 coated SHT04532C tablet, containing 0.451 mg Metafolin (L-5-methyltetrahydrofolate calcium [L-5-MTHF Ca])
Arm/Group | EE 0.02mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE20/DRSP/L-5-MTHF Ca) | L-5-MTHF Ca 0.451 mg (Metafolin)
Number analyzed (Participants) | 39 | 40
nmol·h/L | 214 [195 to 235] | 217 [199 to 237]
Statistical Analysis 1: Comparison: EE 0.02mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE20/DRSP/L-5-MTHF Ca) vs L-5-MTHF Ca 0.451 mg (Metafolin); [analysis description as in outcome 5, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA — The equivalence test was done using a 90% confidence interval, no p-value was to be calculated; mean ratio = 98.16, 90% CI [93.95 to 102.57] — [estimate comment as in outcome 5, analysis 1]

7. Primary Outcome: Mean Maximum Concentration (Cmax) of L-5-methyl-THF (Baseline Uncorrected) Incl. Bioequivalence (BE) Evaluation
Description: The baseline uncorrected Cmax is a measure of the highest measured drug concentration including the endogenous L-5-methyl-THF level. It is obtained by collecting a series of blood samples and measuring the concentrations of L-5-methyl-THF in each sample.
Time Frame: up to 12 hours after administration
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | EE 0.02mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE20/DRSP/L-5-MTHF Ca) | L-5-MTHF Ca 0.451 mg (Metafolin)
Number analyzed (Participants) | 40 | 40
nmol/L | 57.9 [52.6 to 63.6] | 57.7 [51.7 to 64.4]
Statistical Analysis 1: Comparison: EE 0.02mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE20/DRSP/L-5-MTHF Ca) vs L-5-MTHF Ca 0.451 mg (Metafolin); 40 volunteers qualified for statistical analysis of BE and all 40 volunteers with valid concentration time profiles were included in the pharmacokinetic (PK) analysis; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA — The equivalence test was done using a 90% confidence interval, no p-value was to be calculated; mean ratio = 100.28, 90% CI [93.15 to 107.95] — [estimate comment as in outcome 5, analysis 1]

8. Primary Outcome: Mean Area Under the Concentration-time Curve From Administration to the Last Measurement [AUC(0-tlast)] of L-5-methyl-THF (Baseline Uncorrected) Incl. Bioequivalence (BE) Evaluation
Description: The baseline uncorrected AUC is a measure of the systemic drug exposure provided by the treatment including the endogenous L-5-methyl-THF level. It is obtained by collecting a series of blood samples and measuring the concentrations of L-5-methyl-THF in each sample.
Time Frame: up to 12 hours after administration
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: nmol·h/L
Arm/Group | EE 0.02mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE20/DRSP/L-5-MTHF Ca) | L-5-MTHF Ca 0.451 mg (Metafolin)
Number analyzed (Participants) | 40 | 40
nmol·h/L | 370 [333 to 412] | 370 [334 to 411]
Statistical Analysis 1: Comparison: EE 0.02mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE20/DRSP/L-5-MTHF Ca) vs L-5-MTHF Ca 0.451 mg (Metafolin); [analysis description as in outcome 7, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA — The equivalence test was done using a 90% confidence interval, no p-value was to be calculated; mean ratio = 99.88, 90% CI [95.38 to 104.58] — [estimate comment as in outcome 5, analysis 1]

9. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) of EE
Description: Tmax refers to the time after dosing when a drug attains its highest measurable concentration (Cmax). It is obtained by collecting a series of blood samples at various times after dosing, and measuring them for drug content
Time Frame: up to 96 hours after administration
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | EE 0.02 mg/DRSP 3 mg (YAZ, BAY86-5300) | EE 0.02mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE20/DRSP/L-5-MTHF Ca)
Number analyzed (Participants) | 39 | 39
hours | 1.50 [0.50 to 4.00] | 1.52 [1.00 to 4.18]

10. Secondary Outcome: Mean Area Under the Concentration-time Curve From Administration up to 72h AUC(0-72h) of DRSP
Description: as for outcome 2
Time Frame: up to 72 hours after administration
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng·h/mL
Arm/Group | EE 0.02 mg/DRSP 3 mg (YAZ, BAY86-5300) | EE 0.02mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE20/DRSP/L-5-MTHF Ca)
Number analyzed (Participants) | 34 | 36
ng·h/mL | 350 [328 to 373] | 344 [319 to 371]
Statistical Analysis 1: Comparison: EE 0.02 mg/DRSP 3 mg (YAZ, BAY86-5300) vs EE 0.02mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE20/DRSP/L-5-MTHF Ca); 32 volunteers qualified for statistical analysis of BE whereas all 34 (YAZ) and 36 (EE20/DRSP/L-5-MTHF Ca) volunteers with valid concentration time profiles were included in the pharmacokinetic (PK) analysis; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA — The equivalence test was done using a 90% confidence interval, no p-value was to be calculated; mean ratio = 100.30, 90% CI [97.65 to 103.02] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) of DRSP
Description: as for outcome 9
Time Frame: up to 168 hours after administration
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | EE 0.02 mg/DRSP 3 mg (YAZ, BAY86-5300) | EE 0.02mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE20/DRSP/L-5-MTHF Ca)
Number analyzed (Participants) | 35 | 36
hours | 2.00 [0.50 to 4.00] | 2.00 [0.50 to 4.10]

12. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) of L-5-methyl-THF
Description: as for outcome 9
Time Frame: up to 12 hours after administration
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | EE 0.02mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE20/DRSP/L-5-MTHF Ca) | L-5-MTHF Ca 0.451 mg (Metafolin)
Number analyzed (Participants) | 40 | 40
hours | 0.50 [0.00 to 4.00] | 0.50 [0.50 to 2.00]

ADVERSE EVENTS:
Arm/Group | EE 0.02 mg/DRSP 3 mg (YAZ, BAY86-5300) | EE 0.02mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE20/DRSP/L-5-MTHF Ca) | L-5-MTHF Ca 0.451 mg (Metafolin)
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/41 | 0/43
Other Adverse Events (participants affected / at risk) | 37/43 | 30/41 | 34/43
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EE 0.02 mg/DRSP 3 mg (YAZ, BAY86-5300) (N=43) | EE 0.02mg/DRSP 3mg/L-5-MTHF Ca 0.451mg (EE20/DRSP/L-5-MTHF Ca) (N=41) | L-5-MTHF Ca 0.451 mg (Metafolin) (N=43)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eyelid irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 4 (4) | 2 (2) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 4 (4) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 5 (5) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 11 (11) | 5 (5)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (4) | 2 (2)
Asthenia (General disorders) | 4 (4) | 0 (0) | 0 (0)
Catheter site haematoma (General disorders) | 0 (0) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 3 (3) | 0 (0)
Catheter site related reaction (General disorders) | 2 (3) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (3) | 0 (0)
Discomfort (General disorders) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 5 (6) | 5 (6) | 2 (2)
Feeling cold (General disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic intolerance (General disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral coldness (General disorders) | 2 (2) | 0 (0) | 0 (0)
Puncture site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Thirst (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Blepharospasm (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 3 (3)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Serum ferritin decreased (Investigations) | 7 (7) | 6 (6) | 8 (8)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (4) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 15 (17) | 9 (11) | 11 (13)
Hypoaesthesia (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0)
Syncope vasovagal (Nervous system disorders) | 7 (8) | 3 (4) | 2 (2)
Tremor (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Emotional disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 10 (10) | 9 (9) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dental treatment (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI (principal investigator) of CRO (contract research organization) will refrain from publishing any data or information generated or derived as a result of the performance of the Services.